CLINICAL TRIAL: NCT04433000
Title: Comparison Between a Pocket Sized and a High End Ultrasound Scanner in the Evaluation of Lung Involvement in Patients With Covid-19 Pneumonia
Brief Title: Reliability of a Pocket Sized Ultrasound Scanner in the Evaluation Covid-19 Pneumonia
Acronym: USCovid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Piersante Sestini, Associate professor of respiratory diseases, University of Siena
Other Study IDs: USCovid
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Covid-19 Pneumonia
Keywords: Covid-19; pneumonia; lung ultrasound
MeSH Terms: conditions — COVID-19; Pneumonia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Butterfly — Standardized lung ultrasound scan with two different instruments
  Other Names: GE Healthcare Venue GO

SUMMARY:
Ultrasound imaging of the lung (LUS) and associated tissues has demonstrated clinical utility in COVID-19 patients. The aim of the present study was to evaluate the possibilities of a portable pocket-sized ultrasound scanner in the evaluation of lung involvement in patients with COVID-19 pneumonia, in comparison with a high end ultrasound scanner.

Statisical analysis will be performed with Stata for Windows V 16 (Stata corp, Texas College, TX). Power size estimation using Medcalc 19.3.1, (MedCalc Software Ltd, Ostenda, B) showed that hat 34 patients would be required for the comparison of the two methods using the Bland-Altman method assuming a mean difference in total score of 1±1, a false positive rate (α) of 0.05 and a false negative rate of 0.1 (β=0.9).

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19), caused by infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), emerged in China in December 2019 and quickly spread all over the globe. The clinical features are fever, dyspnoea, dry cough, fatigue and diarrhoea (1). Pharyngodynia, nasal congestion, rhinorrhoea and anosmia have also been reported . Interstitial pneumonia is very common and a high percentage of patients (9-11%) develop severe acute respiratory distress syndrome (ARDS) and require intensive care. Current therapeutic strategy involves agents counteracting viral invasion and replication, and inhibitors of cytokine-sustained inflammatory reactions. No specific antiviral therapy has yet been identified.

Ultrasound imaging of the lung (LUS) and associated tissues has demonstrated clinical utility in COVID-19 patients, due to the typical sonographic characteristics of affected lungs. It provides indications for clinical decisions and the management of associated respiratory failure and lung injury.

The aim of the present study was to evaluate the possibilities of a portable pocket-sized ultrasound scanner in the evaluation of lung involvement in patients with COVID-19 pneumonia.

We will perform 34 LUS (lung ultrasound scan) evaluations on patients admitted to the COVID Unit of Siena University Hospital with symptoms compatible with COVID-19, a positive SARS-CoV-2 nasal-pharyngeal swab and radiological evidence of interstitial pneumonia.

The patients will be divided into three severity categories based on respiratory impairment: Mild PaO2/FiO2 > 300 in room air or oxygen flow; Moderate PaO2/FiO2 between 150 and 300 in room air or oxygen-therapy, CPAP, NIV or HFNC; Severe PaO2/FiO2 < 150 on oxygen-therapy, CPAP, NIV, HFNC or mechanical ventilation.

The lung ultrasound scans will be performed on the same day with a standard ultrasound scanner (GE Healthcare, Venue GO) and a pocket-sized ultrasound scanner (Butterfly Network Inc., Butterfly iQ) for clinical purposes; lung preset will be used with both scanners. Up to six regions of the chest will be identified: anterosuperior (A); anteroinferior (B); lateralsuperior (C); lateralinferior (D); posterosuperior (E); posteroinferior (F). One of four different aeration patterns will be recorded according to a specific scoring system: A = 0 points (normal aeration, presence of lung sliding with A lines or less than two isolated B lines), B1 = 1 point (moderate loss of lung aeration, multiple well-defined B lines), B2 = 2 points (severe loss of lung aeration, multiple coalescent B lines), C = 3 points (lung consolidation and tissue-like pattern). Pleural effusion and pneumothorax were also recorded. A score of 0 was normal and 36 was the worst. Due to clinical conditions, the upper posterior region (E) could not be explored in some patients, so the mean of the regions explored will be calculated for the purposes of statistical analysis (total sum (0 to 36) divided by number of regions explored (5 or 6 on each side).

ELIGIBILITY:
Inclusion Criteria:

* Admitted to hospital ward with a diagnosis of Covid-19 preumonia, confirmed by a positive rtPCR swab and radiography

Exclusion Criteria:

* Unable/unwilling to cooperate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to hospital ward with a diagnosis of Covid-19 preumonia, confirmed by a positive rtPCR swab and radiography
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Estimated)

PRIMARY OUTCOMES:
Bland-Altman estimate of bias and Limits of Agreement (LoA) of patient mean scores obtained with the two instruments | 1 day
  The more widely accepted measure of agreement beteen two instruments. Bland JM, Altman DG (1986) Statistical method for assessing agreement between two methods of clinical measurement. The Lancet i:307-310

CONTACTS AND LOCATIONS:
Overall Officials: David Bennett, MD, Principal Investigator — Azienda Ospedaliera Universitaria Senese
Locations (1):
- Azienda Ospedaliera Universitaria Senese, Siena, Si, Italy

IPD SHARING:
Plan to Share IPD: Yes
The whole anonymized dataset could be shared
Supporting Information: Study Protocol
Time Frame: from the month of July, for one year
Access Criteria: on request by email